CLINICAL TRIAL: NCT07190040
Title: Integrating Multi-Omics Data for Enhanced Prognosis Prediction in Gastric Cancer Post-Neoadjuvant Therapy
Status: Completed | Type: Observational
Sponsor: Chang-Ming Huang, Prof. (Other)
Responsible Party: Sponsor-Investigator, Chang-Ming Huang, Prof., Prof., Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: 2025NAT01
Record Dates: First submitted 2025-09-13; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Gastric Cancer (GC)
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Study Protocol: Integrating Multi-Omics Data for Prognosis Prediction in Gastric Cancer Post-Neoadjuvant Therapy

Objective:

To develop and validate an integrative prognostic nomogram for patients with locally advanced gastric cancer (LAGC) undergoing neoadjuvant therapy, combining deep learning-derived radiomic features (DeepScore), transcriptome-based immune scores (ImmuneScore), and ypTNM staging.

Study Design:

A retrospective, single-center cohort study.

Participants:

A total of 179 LAGC patients who received neoadjuvant therapy followed by radical gastrectomy at Fujian Medical University Union Hospital between January 2019 and December 2022. Patients were divided into a training cohort (n = 125) and an independent validation cohort (n = 54).

Data Collection:

Baseline contrast-enhanced CT scans prior to neoadjuvant therapy were used for radiomic analysis. Postoperative tumor RNA sequencing data were used for immune profiling. Clinical and pathological data, including ypTNM stage, were collected from medical records.

Methods:

DeepScore: Extracted from CT images using a ResNet18-based deep learning model. Significant features were selected via univariate Cox and LASSO regression.

ImmuneScore: Calculated from RNA-seq data using the ESTIMATE algorithm to assess tumor immune infiltration.

Nomogram Construction: A multi-omics nomogram was developed using multivariate Cox regression incorporating DeepScore, ImmuneScore, and ypTNM stage.

Validation: Model performance was evaluated using time-dependent ROC analysis (AUC) and Kaplan-Meier survival analysis with log-rank tests in both cohorts.

Primary Outcomes:

Disease-free survival (DFS) and overall survival (OS).

Statistical Analysis:

Survival analyses were performed using Kaplan-Meier and Cox regression models. AUC values were computed for 1-, 2-, and 3-year DFS predictions. All analyses were conducted in R (v4.4.3).

ELIGIBILITY:
Inclusion Criteria:

* Gastric adenocarcinoma confirmed pathologically via gastroscopy;
* Clinical staging of cT3/T4N0/+M0 with a history of receiving at least two cycles of neoadjuvant therapy
* No prior history of other malignant tumors
* Completion of radical gastrectomy

Exclusion Criteria:

* Gastric cancer originating from the remnant stomach
* Absence of baseline computed tomography (CT) data prior to treatment or suboptimal CT image quality that could compromise the accuracy of radiomic information extraction
* Absence of postoperative transcriptome data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with locally advanced gastric cancer who underwent neoadjuvant therapy
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
the Area Under the Curve | 2023.01.31-2025.05.31
  The model's predictive accuracy was evaluated by computing the Area Under the Curve for predicting 1-year, 2-year, and 3-year disease-free survival.

SECONDARY OUTCOMES:
Disease-free survival | 2023.01.31-2025.05.31
  The log-rank test was utilized to compare disease-free survival and overall survival curves between these groups.

OTHER OUTCOMES:
Overall survival | 2023.01.31-2025.05.31
  The log-rank test was utilized to compare disease-free survival and overall survival curves between these groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China